CLINICAL TRIAL: NCT03933150
Title: Caudal Epidural Steroid Injection Ultrasound Guided Versus Fluoroscopy Guided in Treatment of Refractory Lumbar Disc Prolapse With Radiculopathy
Brief Title: Caudal Epidural Steroid Injection Ultrasound Guided in LDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: code: MS/16.06.46.
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2019-05

CONDITIONS: Refractory Lumbar Disc Prolapse
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Type of randomization:
  Patients were randomly divided into 2 treatment groups. For allotting, bunches bits of paper were set up in a similar number of patients. The name of treatment strategies was composed on the bits of paper. At that point, patients were made a request to take one paper and this is the treatment sort for every individual was determined.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasoun guided caudal epidural injection (Other): A. Ultrasound-Guided CESI (Group 1) All the injection procedures were performed as an outpatient clinic setting. We used Acuson P300 (Siemens, Italy) with a linear transducer at 6 to 12 MHz as the US instrument, another curved transducer at 2-5 MHz was available for obese patients.
  Interventions: Device: ultrasound guided caudal epidural injection
- fluoroscopy guided caudal epidural injection (Other): B. Fluoroscopy-Guided CESI (Group 2) All the injection procedures were performed in a specialized room with a FL device in the radiology department. We used a FL device GS 1004 with ALLURA XPER FD 20 system (Philips, Holland) with X-ray tube housing assembly, X-ray tube, beam limiting device and image receptor
  Interventions: Device: ultrasound guided caudal epidural injection

INTERVENTIONS:
Device: ultrasound guided caudal epidural injection — A. Ultrasound-Guided CESI (Group 1) All the injection procedures were performed as an outpatient clinic setting. We used Acuson P300 (Siemens, Italy) with a linear transducer at 6 to 12 MHz as the US instrument, another curved transducer at 2-5 MHz was available for obese patients.
  B. Fluoroscopy-Guided CESI (Group 2) All the injection procedures were performed in a specialized room with a FL device in the radiology department. We used a FL device GS 1004 with ALLURA XPER FD 20 system (Philips, Holland) with X-ray tube housing assembly, X-ray tube, beam limiting device and image receptor
  Other Names: fluoroscopy guided caudal epidural injection

SUMMARY:
Patients with LDP with unilateral radiculopathy diagnosed by routine clinical examination and MRI, in whom conservative treatment (medical treatment and physiotherapy) failed for more than 6 weeks and refuse surgery or were unfit for surgery A. Ultrasound-Guided CESI (Group 1) All the injection procedures were performed as an outpatient clinic setting. We used Acuson P300 (Siemens, Italy) with a linear transducer at 6 to 12 MHz as the US instrument, another curved transducer at 2-5 MHz was available for obese patients.

All the injection procedures were performed in a specialized room with a FL device in the radiology department. We used a FL device GS 1004 with ALLURA XPER FD 20 system (Philips, Holland) with X-ray tube housing assembly, X-ray tube, beam limiting device and image receptor

DETAILED DESCRIPTION:
228 patients suffering from LDP with radiculopathy,recruited from the outpatient Clinic of Rheumatology and Rehabilitation department at Mansoura University Hospital were assessed for eligibility to participate in this study.

Those who met the inclusion criteria wereselected. Conversely, those who did not meet inclusion criteria or met the exclusion criteria were excluded.Accordingly, 136 patients who met the inclusion criteria were divided into two groups:

* Group 1: included 68 patients who received US-guided CESI. They were 39 females and 29 males. Their age ranged from 23 to 65.
* Group 2: included 68 patients who received FL-guided CESI. They were 38 females and 30 males. Their age ranged from 22 to 62.

A written consent was obtained from each participant sharing in this study. The institutional research board of faculty of medicine, Mansoura University, approved this study, code: MS/16.06.46.

Inclusion Criteria:

Patients with LDP with unilateral radiculopathy diagnosed by routine clinical examination and MRI, in whom conservative treatment (medical treatment and physiotherapy) failed for more than 6 weeks and refuse surgery or were unfit for surgery

Exclusion Criteria:

Vertebral fractures, direct trauma, spinal inflammatory disease, spinal infection, bleeding tendency, LBP with tumors, bilateral radiculopathy, cauda equina syndrome, spinal canal stenosis, post-laminectomy surgery, diabetic and hypertensive patients.

Study design:

Randomized controlled clinical trial.

Type of randomization:

Patients were randomly divided into 2 treatment groups. For allotting, bunches bits of paper were set up in a similar number of patients. The name of treatment strategies was composed on the bits of paper. At that point, patients were made a request to take one paper and this is the treatment sort for every individual was determined.

I. Clinical Evaluation:

1. History Taking:including

1. Personal history

   o Name, age, sex, occupation, marital status, offspring and smoking.
2. Present History

   * Pain: onset, course, duration, site, nature, radiation and modifying factors.
   * Associated symptoms: fever, unexplained weight loss, night pain, chronic cough, stiffness, pain in other joints, skin lesions, diarrhea, urogenital diseases, eye lesions, anxiety, depression, fatigue or sleep disturbance.
   * Neurological symptoms: numbness, paresthesia, muscle weakness, claudication, or sphincteric disturbance.
   * Articular symptoms : of other joints including cervical, hips and knees
   * Symptoms related to other systems: respiratory, cardiovascular, gastrointestinal, urinary, and gynecological systems.
   * Work related conditions
3. Past History III. Assessment of pain Patients were assessed before treatment, 1 month and 3 months after the injection using VAS.

IV. Assessment of pain and function Patients were assessed before treatment, 1 month and 3 months after the injection procedure by the ODI.

All the eligible patients were treated with either US-guided or FL-guided CESI, were administered a mixture of 20 cc (0.5% lidocaine 18.0 mL &2ml of triamcinolone acetonide 40 mg/1ml) (Bicket, et al., 2015; Manchikanti, et al., 2015b).

A. Ultrasound-Guided CESI (Group 1) All the injection procedures were performed as an outpatient clinic setting. We used Acuson P300 (Siemens, Italy) with a linear transducer at 6 to 12 MHz as the US instrument, another curved transducer at 2-5 MHz was available for obese patients.

B. Fluoroscopy-Guided CESI (Group 2) All the injection procedures were performed in a specialized room with a FL device in the radiology department. We used a FL device GS 1004 with ALLURA XPER FD 20 system (Philips, Holland) with X-ray tube housing assembly, X-ray tube, beam limiting device and image receptor

ELIGIBILITY:
Inclusion Criteria:

- Patients with LDP with unilateral radiculopathy diagnosed by routine clinical examination and MRI,

Exclusion Criteria:

* Vertebral fractures, direct trauma, spinal inflammatory disease, spinal infection, bleeding tendency, LBP with tumors, bilateral radiculopathy, cauda equina syndrome, spinal canal stenosis, post-laminectomy surgery, diabetic and hypertensive patients.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
change of degree of pain from base line Patients were assessed before treatment, 1 month and 3 months after the injection using VAS. | assessed immediately before injection,1 month after injection,3 month after injection
  Visual analog scale for pain is a measurement tool that measures a characteristic or attitude that is believed to range across a continuum of values.It is usually a horizontal line, 100 mm in length, anchored by verbal descriptors at each end: 'no pain' and 'worst pain possible'. The patients place a mark on the line that represented their level of pain intensity. The distance from the left-hand side was measured in millimeters. This distance quantifies pain level. The following cut points on has been suggested: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100mm) (Smeets, et al., 2011; Elfving, et al., 2016).
change of Straight leg raising test (SLRT) (Lasègue's sign from base line | assessed immediately before injection,1 month after injection,3 month after injection
  One of the most common clinical diagnostic tests (Iversen, et al., 2013). The patient lies on a table in supine position. With one hand set over the knee of the leg being examined, the examiner applies enough firm pressureto keep the knee in full extension. With the alternate hand cupped under the heel, the examiner raises the straight limb gradually. Sciatic nerve compression is indicated if pain is agonized or worsened on raising the leg to a level more than 25° but lower than 75º. The ankle is dorsiflexed as the leg is held at the limit of straight-leg raising (onset). Symptoms are exaggerated in persons who have nerve root compression as the reason (De Luigi and Fitzpatrick, 2011).
change of Femoral stretch test from base line | assessed immediately before injection,1 month after injection,3 month after injection
  While patient lies prone, the knee is inactively flexed to the thigh and the hip is pas extended; thetest ispositive if the patient encounters pain in front of the thigh (Magee, 2013).
change of Modified Schober's test from base line | assessed immediately before injection,1 month after injection,3 month after injection
  While the patient is standing erect, marks are made 5 cm below and 10 cm above the lumbosacral junction (dimples of Venus) and the distance between the two marks is measured. Then measurement is repeated with the patient in full forward flexion (Fig. 9). In general, the measure should increase by at least 5 cm to 21 cm. An increase of less than 5 cm advocates decreased lumbar spinal mobility.

SECONDARY OUTCOMES:
change of pain and function from base line: Oswestry Disability Index Patients were assessed before treatment, 1 month and 3 months after the injection procedure by the ODI. | assessed immediately before injection,1 month after injection,3 month after injection
  Oswestry Disability Index (Fairbank and Pynsent, 2000) It is a self-administered questionnaire compromised of 10 sections; each section is scored on a 0-5 scale, 5 representing the greatest disability (see the Appendix).
  It is composed of 10 short-termsectors. The index is calculated by dividing the summed score by the total possible score, after that it is multiplied by 100 and expressed as a percentage. Thus, for the not answered questions, the denominator is reduced by 5 for each.
  Interpretation of scores:
  0% to 20%:minimal disability:The patient can cope with most living activities. Usually no treatment is indicated apart from advice on lifting sitting and exercise.
  21%-40%: moderate disability:The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Mansoura University, Al Mansurah, Dakahlia Provence, Egypt